CLINICAL TRIAL: NCT01039987
Title: Consortium for Radiologic Imaging Studies of Polycystic Kidney Disease (CRISP) II
Brief Title: Consortium for Radiologic Imaging Studies of Polycystic Kidney Disease
Acronym: CRISP II
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kyongtae Ty Bae, M.D., Ph.D., Professor of Radiology and Bioengineering, University of Pittsburgh
Other Study IDs: DK056961
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal dominant polycystic kidney disease; ADPKD; kidney; Biomarker; MRI
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The Division of Kidney Urology and Hematology Disease (DKUHD) of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) funded a cooperative agreement (UO1) for a consortium of participating clinical centers (PCCs) and a data coordinating and imaging analysis center (DCIAC) to develop and implement studies to test whether imaging techniques can provide accurate and reproducible markers of progression of renal disease in patients with polycystic kidney disease.

The awarded participating clinical centers are Emory University, University of Kansas, and Mayo Foundation (with a subcontract to the University of Alabama). The awarded DCIAC is Washington University in St. Louis. Due to the relocation of the DCIAC P.I. from Washington University to the University of Pittsburgh, the DCIAC for CRISP II is located at the University of Pittsburgh.

DETAILED DESCRIPTION:
The goal of the CRISP Study is to conduct a prospective, longitudinal trial to evaluate the accuracy and validity of magnetic resonance imaging to determine disease progression in ADPKD defined as a change in both renal and renal cyst volumes and renal function over time.

ELIGIBILITY:
Inclusion Criteria:

1. CRISP I participants will be invited to participate in CRISP II. At entry into CRISP I participants met a number of inclusion and exclusion criteria.

Exclusion Criteria:

1. Current psychiatric or addiction or non-compliance disorder that in the discretion of the principal investigator indicates that the subject will not successfully complete the study;
2. Current medical problem that in the discretion of the principal investigator would make unsafe the participation in the study;
3. Inability to provide written informed consent

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who are diagnosed with ADPKD between the ages of 15 and 45 with risk factors (2/3 of the study population) or without risk factors (1/3 of the study population)for progression to ESRD with relatively normal renal function were be eligible for recruitment into the CRISP I study. The objective of the recruitment process was to identify ADPKD participants with the appropriate level of renal function who are either at high or low risk for progression to ESRD, who will be available for the entire follow-up period and who are likely to be compliant with the study protocols and visit schedules.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 1999-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
kidney volume | three years

CONTACTS AND LOCATIONS:
Overall Officials: Marva Moxey-Mims, M.D., Study Director — NIH, NIDDK, DKUH; K. Ty BAE, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - University of Kansas, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Bae K, Park B, Sun H, Wang J, Tao C, Chapman AB, Torres VE, Grantham JJ, Mrug M, Bennett WM, Flessner MF, Landsittel DP, Bae KT; Consortium for Radiologic Imaging Studies of Polycystic Kidney Disease (CRISP). Segmentation of individual renal cysts from MR images in patients with autosomal dominant polycystic kidney disease. Clin J Am Soc Nephrol. 2013 Jul;8(7):1089-97. doi: 10.2215/CJN.10561012. Epub 2013 Mar 21. PMID 23520042